CLINICAL TRIAL: NCT04530890
Title: Interest of Circulating Tumor DNA in Digestive and Gynecologic/Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ADIGYN
Record Dates: First submitted 2020-08-11; First posted 2020-08-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Digestive Cancer; Gynecologic Cancer; Circulating Tumor DNA; Exosomes
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm only (Experimental): Only one arm with blood samples
  Interventions: Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Blood samples — Only blood samples at different times of treatment

SUMMARY:
Circulating tumor DNA (ctDNA) offers the possibility of accessing the tumor genome from circulating blood through a simple blood test. It is currently used for diagnostic, prognostic and predictive purposes of response or resistance to oncological treatments. These advances in ctDNA have been made possible by major developments in molecular biology techniques in recent years, as the detection of ctDNA requires very sensitive techniques such as Next Generation Sequencing (NGS).

CtDNA overcomes this problem of very limiting tumor heterogeneity during a solid biopsy. All of these applications make circulating DNA an increasingly essential tool in the management of cancer patients. The studies are currently in most cases on small numbers and are retrospective.

In addition, exosomes are also a biomarker of the future that can also be detected in the bloodstream . Exosomes are nanovesicles 50 to 200 nm in diameter released into the extracellular environment via the endosomal pathway by fusion with the plasma membrane. They are very informative since they transport tumor genetic material in the form of DNA, mRNA and miRNA, but also adhesion proteins, immunostimulatory molecules and cytoskeleton, enzymes and Heats shock proteins ( HSP).

The aim of the ADIGYN study is to set up a large prospective cohort to assess the diagnostic, prognostic and predictive impact of ctDNA and exosomes in digestive and gynecological / breast cancers. From the circulating DNA, we characterize the ActDNA on the molecular level thanks to the study of different point mutations usually used but also of new described mutations having a therapeutic impact and the search for other genetic alterations having an impact on the therapeutic strategy (such as microsatellite instability) or the study of exosomes and their composition. To assess resistance to oncological treatments, ctDNA will be analyzed at the start of treatment, during treatment, during progression and / or relapse and also during monitoring or treatment break

ELIGIBILITY:
Inclusion Criteria:

* Digestive or gynecological / breast cancer proven or suspected, requiring oncological treatment (chemotherapy or immunotherapy)
* Major patient
* Patients benefiting from a Social Security scheme or benefiting through the intermediary of a third party
* Information note and collection of non-opposition after clear and fair information about the study

Exclusion Criteria:

* Linguistic or psychological refusal or inability to understand and / or sign the information and no-objection note
* History of a cancer other than that allowing inclusion in the 5 years preceding inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
To assess the prognostic impact of ctDNA (mortality) in digestive and gynecological / breast cancers. | Through study completion, an average of 12 months
  Correlation between ctDNA and overall survival

SECONDARY OUTCOMES:
Evaluate the diagnostic value of ctDNA and exosomes | Through study completion, an average of 12 months
  ct DNA and exosomes analyses can be new tools for cancer diagnosis
Evaluate the prognostic impact of exosomes and their composition | Through study completion, an average of 12 months
  There are many kind of exomossomes with few different composition and different roles
Evaluate the predictive benefit of response / resistance to ctDNA and exosome treatments | Through study completion, an average of 12 months
  Correkation between ctDNA/exosomes and progression free survival
Evaluate the possibility of detecting certain molecular alterations using ctDNA and exosomes | Through study completion, an average of 12 months
  With new technics of biology molecular, we are going to try to detect molecular alterations in ctDNA /exosomes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU POitiers, Poitiers, France